CLINICAL TRIAL: NCT03102216
Title: An Assessment of the Impact of Enhanced Workflow Patterns Associated With Upfront, Early Point-of-care Testing on Costs, Waiting and Disposition Times in an Emergency Department
Brief Title: Early Point-Of-Care Blood Tests, ECG & X-rays in the Emergency Department
Acronym: EPOC-BEX-ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helen Joseph Hospital (Other)
Collaborators: Abbott Point of Care (Industry); University of Johannesburg (Other); Lodox Systems (Ltd) (Unknown)
Responsible Party: Principal Investigator, Dr LN Goldstein, Head: Department of Emergency Medicine, Helen Joseph Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EPOC-BEX-ED
Record Dates: First submitted 2017-03-16; First posted 2017-04-05 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Emergency Medicine; Point-of-Care Testing
MeSH Terms: interventions — Electrocardiography

STUDY DESIGN:
Intervention Model Description: Investigator-initiated, Prospective, Randomised, Control Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Current workflow pathway (No Intervention): In the Current (normal) Workflow Pathway, after a patient is triaged, they are reviewed by the doctor. It is routine for the doctor to then order diagnostic tests/investigations that include blood tests, which are analysed at the laboratory, x-rays, which are performed in the Radiology department, and an ECG, which is performed by an ECG technician. Once the results of those tests are ready, the doctor will then review the patient a second time with all the results. The decision for patient disposition will then be made
- Enhanced workflow pathway iSTAT (Experimental): Patients will receive i-STAT point-of-care troponin, INR (International Normalised Ratio), CG4(blood gas analysis) and chem8 tests prior to seeing the doctor.
  Interventions: Diagnostic Test: iSTAT
- Enhanced workflow pathway iSTAT CBC (Experimental): Patients will receive iSTAT point-of-care troponin, INR, CG4+ and chem8 tests as well as a CBC prior to seeing the doctor.
  Interventions: Diagnostic Test: iSTAT; Diagnostic Test: CBC
- Enhanced workflow pathway ECG (Experimental): Patients will receive a 12lead, v1R-v6R(right sided ECG leads) and V7-V9 ECG prior to seeing the doctor.
  Interventions: Diagnostic Test: ECG
- Enhanced workflow pathway Lodox (Experimental): Patients will receive a supine AP and lateral lodox (low dose x-ray) of their chest and abdomen prior to seeing the doctor.
  Interventions: Diagnostic Test: Lodox
- Enhanced workflow pathway iSTAT ECG (Experimental): Patients will receive iSTAT point-of-care troponin, INR, CG4+ and chem8 tests as well as 12lead, v1R-v6R and V7-V9 ECG prior to seeing the doctor.
  Interventions: Diagnostic Test: iSTAT; Diagnostic Test: ECG
- Enhanced workflow pathway iSTAT, CBC ECG (Experimental): Patients will receive iSTAT point-of-care troponin, INR, CG4+ and chem8 tests, CBC and 12lead, v1R-v6R and V7-V9 ECG prior to seeing the doctor.
  Interventions: Diagnostic Test: iSTAT; Diagnostic Test: CBC; Diagnostic Test: ECG
- Enhanced workflow pathway iSTAT lodox (Experimental): Patients will receive iSTAT point-of-care troponin, INR, CG4+ and chem8 tests and Lodox prior to seeing the doctor.
  Interventions: Diagnostic Test: iSTAT; Diagnostic Test: Lodox
- Enhanced workflow pathway iSTAT CBC Lodox (Experimental): iSTAT point-of-care troponin, INR, CG4+ and chem8 tests; CBC and Lodox prior to seeing the doctor.
  Interventions: Diagnostic Test: iSTAT; Diagnostic Test: CBC; Diagnostic Test: Lodox
- Enhanced workflow pathway ECG Lodox (Experimental): Patients will receive LODOX and 12lead, v1R-v6R and V7-V9 ECG prior to seeing the doctor.
  Interventions: Diagnostic Test: ECG; Diagnostic Test: Lodox
- Enhanced workflow pathway iSTAT ECG Lodox (Experimental): iSTAT point-of-care troponin, INR, CG4+ and chem8 tests; LODOX and 12lead, v1R-v6R and V7-V9 ECG prior to seeing the doctor
  Interventions: Diagnostic Test: iSTAT; Diagnostic Test: ECG; Diagnostic Test: Lodox
- Enhanced workflow pathway iSTAT CBC ECG Lodox (Experimental): Patients will receive iSTAT point-of-care troponin, INR, CG4+ and chem8 tests; CBC, LODOX and 12lead, v1R-v6R and V7-V9 ECG prior to seeing the doctor.
  Interventions: Diagnostic Test: iSTAT; Diagnostic Test: CBC; Diagnostic Test: ECG; Diagnostic Test: Lodox

INTERVENTIONS:
Diagnostic Test: iSTAT — iSTAT troponin, INR, CG4+ and Chem8
  Arms: Enhanced workflow pathway iSTAT; Enhanced workflow pathway iSTAT CBC; Enhanced workflow pathway iSTAT CBC ECG Lodox; Enhanced workflow pathway iSTAT CBC Lodox; Enhanced workflow pathway iSTAT ECG; Enhanced workflow pathway iSTAT ECG Lodox; Enhanced workflow pathway iSTAT lodox; Enhanced workflow pathway iSTAT, CBC ECG
Diagnostic Test: CBC — Complete Blood Count
  Arms: Enhanced workflow pathway iSTAT CBC; Enhanced workflow pathway iSTAT CBC ECG Lodox; Enhanced workflow pathway iSTAT CBC Lodox; Enhanced workflow pathway iSTAT, CBC ECG
Diagnostic Test: ECG — ElectroCardioGram
  Arms: Enhanced workflow pathway ECG; Enhanced workflow pathway ECG Lodox; Enhanced workflow pathway iSTAT CBC ECG Lodox; Enhanced workflow pathway iSTAT ECG; Enhanced workflow pathway iSTAT ECG Lodox; Enhanced workflow pathway iSTAT, CBC ECG
Diagnostic Test: Lodox — Low dose x-ray
  Arms: Enhanced workflow pathway ECG Lodox; Enhanced workflow pathway Lodox; Enhanced workflow pathway iSTAT CBC ECG Lodox; Enhanced workflow pathway iSTAT CBC Lodox; Enhanced workflow pathway iSTAT ECG Lodox; Enhanced workflow pathway iSTAT lodox

SUMMARY:
The 2015 Abbott Point-of-Care Great Minds Summit in Berlin presented novel research that showed the potential for upfront, point-of-care (POC) blood testing to improve waiting times, costs and patient flow in the Emergency Department (ED). POC testing has become a focus area for enquiry as EDs worldwide look for ways to cope with over-crowding and reduce waiting times.

In South African EDs, the target time for patients to be seen is dictated by their triage category. Patients triaged Red (critical) should ideally be seen immediately, Orange within 10 minutes, Yellow within 1 hour and Green within 4 hours of arrival. Whilst patients may initially be evaluated within the above time frames, there may be delays in their final disposition due to time lags in obtaining results from special tests and/or investigations. Traditionally, blood tests and other special investigations such as electrocardiograms (ECG) and radiological investigations (x-rays) take place after the doctor has evaluated the patient. Patients (and doctors) then have to wait for the results of these tests before a decision can be made regarding the patient's final disposition.

Instead of sending blood specimens to the laboratory for analysis, POC blood testing refers to selected tests which can be performed in the ED and provide immediate on-site results and thus have the potential to expedite patient management decisions. Similarly, low dose x-ray (LODOX®) is the radiological equivalent of a POC blood test providing a full body x-ray within 19 seconds. LODOX has been evaluated in trauma patients previously but its application as a screening tool for non-trauma patients in the ED has not been properly explored thus far. Electrocardiograms (ECGs) are commonly used in clinical medicine as a POC test to evaluate the heart. Locally, Helen Joseph Hospital ED in Johannesburg has a constant influx of critically ill and injured patients 24 hours a day. The aim of this investigator-initiated, prospective, randomised control trial is to compare and assess the standard workflow pathway currently in use in the ED to a modified pathway that makes use of upfront, early POC tests (blood tests, ECG and/or LODOX) to see if the use of such has any significant effect on costs, waiting times and associated patient flow patterns in the ED.

DETAILED DESCRIPTION:
The Helen Joseph Hospital ED has a constant influx of critically ill and injured patients 24 hours a day. On average, 170 - 200 patients are triaged and evaluated per day - approximately 60 000-70000 patients per annum.

EDs world-wide are constantly looking for ways to decrease patient over-crowding and waiting times. Suggested solutions have included the hiring of additional personnel, creating observation units, ambulance diversion and triage. Some have even tried to improve patient flow by placing a senior consultant in the triage area.

In South African EDs, the South African Triage Scale (SATS) is utilised to assess severity and acuity of patients presenting to the ED. The target time for patients to be seen is dictated by their triage category. Patients triaged Red should ideally be seen immediately, Orange within 10 minutes, Yellow within 1 hour and Green within 4 hours of arrival. Whilst patients may initially be evaluated within these time frames, there may be delays in their final disposition due to time lags in obtaining results from special investigations.

Traditionally, investigations in the ED take place after the doctor has evaluated the patient. Patients (and doctors) then have to wait for the results of the investigations. Further decisions on the patients' ultimate disposition (i.e. either discharged home or admitted for inpatient care) are thus contingent upon the results of the investigations.

POC blood testing (as opposed to sending blood to the laboratory to be analysed) has been shown to be accurate and assist in expediting patient management by decreasing the turnaround time for results. Low dose x-ray (LODOX®) has been marketed as a quick and easy radiological screening tool for trauma patients that can even be used as a triage tool. The LODOX can produce a full body antero-posterior x-ray image within 19 seconds. It is much quicker and exposes the patient to less radiation than a standard radiograph/x-ray. It can therefore also be categorised as the x-ray equivalent of a POC test. Its use has never been evaluated as a tool for non-trauma patients in the ED. Electrocardiograms (ECGs) are commonly used in clinical medicine as a POC test to evaluate the heart.

The aim of this study is therefore to assess whether, individually or in combination, upfront, early POC blood tests, ECGs and/or LODOX can decrease waiting times, reduce costs and improve patient flow in the ED.

ELIGIBILITY:
Inclusion Criteria:

All consenting adult patients older than 18 years old, with the one of the symptom groups below, that present to Helen Joseph Hospital ED, who do not require immediate resuscitation i.e. not triaged red. This will be performed during weekdays only.

Presenting symptom groups:

* Abdominal/epigastric/stomach pain/vomiting
* Psychosis/aggression/hallucinations (see Ethical Considerations)
* Shortness of breath/dyspnoea/cough/chest pain/syncope
* General body pain/weakness
* Overdose

Exclusion Criteria:

* Failure to obtain consent
* Pregnant patients
* Patients who require immediate resuscitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1134 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Decrease waiting and disposition times for patients presenting to the Emergency Department | From patient Arrival in the Emergency Department until disposition (i.e. until the decision to admit or discharge the patient is made) through study completion (approximately 4 months)
  Measurement of waiting and workflow times compared to current workflow pathway

SECONDARY OUTCOMES:
Decrease the costs of special investigations for patients presenting to the Emergency Department | Compare the costs for standard care to costs of point-of-care intervention through study completion (approximately 4 months)
  Measurement of cost implications

CONTACTS AND LOCATIONS:
Locations (1):
- Helen Joseph Hospital Emergency Department, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Altman DG, Bland JM. How to randomise. BMJ. 1999 Sep 11;319(7211):703-4. doi: 10.1136/bmj.319.7211.703. No abstract available. PMID 10480833
- [Result] Hoot NR, Aronsky D. Systematic review of emergency department crowding: causes, effects, and solutions. Ann Emerg Med. 2008 Aug;52(2):126-36. doi: 10.1016/j.annemergmed.2008.03.014. Epub 2008 Apr 23. PMID 18433933
- [Result] Jarvis P, Davies T, Mitchell K, Taylor I, Baker M. Does rapid assessment shorten the amount of time patients spend in the emergency department? Br J Hosp Med (Lond). 2014 Nov;75(11):648-51. doi: 10.12968/hmed.2014.75.11.648. PMID 25383437
- [Result] Stotler BA, Kratz A. Analytical and clinical performance of the epoc blood analysis system: experience at a large tertiary academic medical center. Am J Clin Pathol. 2013 Nov;140(5):715-20. doi: 10.1309/AJCP7QB3QQIBZPEK. PMID 24124152
- [Result] Terris J, Leman P, O'Connor N, Wood R. Making an IMPACT on emergency department flow: improving patient processing assisted by consultant at triage. Emerg Med J. 2004 Sep;21(5):537-41. doi: 10.1136/emj.2002.003913. PMID 15333523
- [Result] Whiley SP, Alves H, Grace S. Full-body x-ray imaging to facilitate triage: a potential aid in high-volume emergency departments. Emerg Med Int. 2013;2013:437078. doi: 10.1155/2013/437078. Epub 2013 Sep 24. PMID 24205438
- [Derived] Goldstein LN, Wells M, Vincent-Lambert C. The cost-effectiveness of upfront point-of-care testing in the emergency department: a secondary analysis of a randomised, controlled trial. Scand J Trauma Resusc Emerg Med. 2019 Dec 11;27(1):110. doi: 10.1186/s13049-019-0687-2. PMID 31829227